CLINICAL TRIAL: NCT05986123
Title: Safety and Efficacy of Topical Cream Containing Natural Plant Extracts, Niacinamide, and Arbutin for Post-inflammatory Hyperpigmentation Skin Among Malaysians
Brief Title: Safety and Efficacy of Topical Cream for Post-inflammatory Hyperpigmentation Skin Among Malaysians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMRAMREC002-23
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Aesthetic; Cosmetic; Post-inflammatory hyperpigmentation (PIH)
MeSH Terms: conditions — Hyperpigmentation | interventions — Prolactin Release-Inhibiting Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical cream for PIH (Other): The topical cream contain combination of niacinamide, arbutin, Scutellaria Baicalensis Root Extract, Centella Asiatica Extract and Camellia Sinensis Leaf Extract.
  Interventions: Other: Topical cream Z for PIH

INTERVENTIONS:
Other: Topical cream Z for PIH — The topical cream Z contain combination of niacinamide, arbutin, Scutellaria Baicalensis Root Extract, Centella Asiatica Extract and Camellia Sinensis Leaf Extract. Participants will used the topical cream twice daily for 20 weeks

SUMMARY:
This study was conducted to determine safety and efficacy of topically applied cream containing combination of niacinamide, arbutin, Scutellaria Baicalensis Root Extract, Centella Asiatica Extract and Camellia Sinensis Leaf Extract for its skin brightening effect on post-inflammatory hyperpigmentation among the Malaysian population. The study duration is 20 weeks and the skin assessment will be carried out at baseline, week 4, week 8, week 12, week 16 and week 20.The main questions this study aims to answer are:

1. To determine the efficacy of topical cream containing natural plant extracts, niacinamide, and arbutin for post-inflammatory hyperpigmentation among Malaysians.
2. To investigate the safety of topical cream containing natural plant extracts, niacinamide, and arbutin for post-inflammatory hyperpigmentation among Malaysians.
3. To assess the participants satisfaction of using topical cream containing natural plant extracts, niacinamide, and arbutin for post-inflammatory hyperpigmentation among Malaysians.

ELIGIBILITY:
Inclusion Criteria:

* Malaysia citizen
* Healthy adult, aged between 18 to 40 years old.
* Participants who have post-inflammatory hyperpigmentation on skin

Exclusion Criteria:

* Participants with skin disorders such as skin infection or skin inflammation.
* Participants who have undergone any skin and cosmetic treatments such as dermal fillers, botox, laser, chemical peels within the last 3 months.
* Participant who is taking isotretinoin for the past 6 or 12 months and immunocompromised patients.
* Pregnant, breastfeeding women or planned for pregnancy during the study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in skin spot level | Baseline, week 4, week 8, week 12, week 16 and week 20.
  Skin spot will be assessed using JANUS III skin analyzer.
Change in hyperpigmentation score | Baseline, week 4, week 8, week 12, week 16 and week 20.
  The hyperpigmented skin area will be assessed based on Modified Melasma Area and Severity Index (mMASI) Score. Scoring system of mMASI score: A, Area of involvement is rated from 0 to 6: (0 indicates absent, 1=<10%, 2= 10% to 90%, 3= 30%-49%, 4= 50%-69%, 5= 70% to 89%, 6=90% to 100%). D, Darkness is rated from 0 to 4: 0= absent, 1=slight hyperpigmentation, 2= mild hyperpigmentation, 3= marked hyperpigmentation, 4=severe hyperpigmentation. Total mMASI score range is 0 (clear) to 24 (most severe melasma) and calculated by adding scores (A and D) for 4 areas of the face. The formula for mMASI score = 0.3×A(forehead)×D (forehead)+0.3×A (left malar) ×D (left malar) + 0.3×A(right malar)×D (right malar)+0.1×A(chin)×D (chin).
Adverse effect after using the topical cream. | Week 20
  Based on adverse effect occurrence on participants that occur during study period (20 weeks)

SECONDARY OUTCOMES:
Participant satisfaction after using the topical cream for 20 weeks. | Week 20
  Participation satisfaction will be evaluated using the Physician Global Assessment (PGA) survey. The subjective score of changes in skin conditions including skin wrinkles, dryness, smoothness, moisturizing and brightening effect will be graded as follows: very satisfied, satisfied, neutral, dissatisfied, very dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No